CLINICAL TRIAL: NCT06461988
Title: An Open-Label, Non-Randomized, Phase II Study to Study the Efficacy of Talquetamab (JNJ-64407564) and Lenalidomide as Post Stem Cell Transplant Maintenance in Multiple Myeloma (OPTIMMAL)
Brief Title: Talquetamab & Lenalidomide as Post Stem Cell Transplant Maintenance in Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-73317; NCI-2024-06734 (Registry Identifier: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma; Post Stem Cell Transplant
Keywords: Talequetamab; Lenalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — talquetamab; Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Talquetamab (Experimental): Study participants will receive talquetamab (JNJ-64407564) for one cycle and a combination of talquetamab and lenalidomide for cycles 2-13 after autologous stem cell transplant (ASCT).
  Interventions: Drug: Talquetamab; Drug: Talquetamab and Lenalidomide

INTERVENTIONS:
Drug: Talquetamab — Talquetamab Step up dosing:
  C1D1: 10 mcg/kg C1D3: 60 mcg/kg C1D5: 400 mcg/kg C1D15: 800 mcg/kg
  Talquetamab 800 mg/kg SC Q4W in 28-day cycle for Cycles 2-13
Drug: Talquetamab and Lenalidomide — Lenalidomide 10 mg, 3 weeks on 1 week off, until PD/ intolerance, C2-13 (Lenalidomide 5 mg for creatinine clearance 30-60 ml/min)

SUMMARY:
Multiple myeloma (MM) is a heterogenous plasma cell malignancy characterized by clonal proliferation of plasma cells and organ damage. Autologous transplantation with high dose chemotherapy is the standard of care in frontline treatment of eligible patients with MM.

DETAILED DESCRIPTION:
This is a phase 2 study to evaluate the efficacy of talquetamab with a combination of lenalidomide, and to determine the safety and longitudinal patient reported symptoms and quality of life.

Twenty participants with MM who plan to undergo or who have undergone autologous stem cell transplant as a part of their initial therapy and meet the eligibility criteria will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have had a confirmed diagnosis of symptomatic multiple myeloma according to according to IMWG diagnostic criteria.
2. Measurable disease at the time of myeloma diagnosis Measurable disease is defined as measurable M protein in the serum (≥ 0.5g/dL) or urine (≥ 200 mg/24h) or serum free light chain assay (defined as dFLC ≥ 10 mg/dL [≥ 100 mg/L]; difference between involved and uninvolved free light chain) at the time of diagnosis. Participants with smoldering myeloma are not eligible until they have progressed to symptomatic myeloma. Participants with purely non-secretory MM at the time of diagnosis as measured by electrophoresis and immunofixation and the absence of Bence Jones proteins in the urine are not eligible.
3. Age >18 years.
4. Patients who have already received transplant should have undergone autologous stem cell transplant with Melphalan 140 mg/m2 within 12 months of start of induction therapy of multiple myeloma and are within day +60-120 post-transplant. Patients who have not already received transplant must have begun induction therapy within 12 months prior to the planned date of transplant.
5. Participants must not be refractory to lenalidomide
6. Participants must not have progressive disease at any time prior to registration
7. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
8. Have clinical laboratory values meeting the following criteria during the Screening Phase and also at start of administration of study treatment:

   - Hemoglobin: ≥ 8 g/dL (≥ 4.96 mmol/L; without transfusion support or erythropoietin use within 7 days before the laboratory test)

   - Platelets: ≥ 75×109/L in participants in whom <50% of bone marrow nucleated cells are plasma cells and ≥ 50×109/L in participants in whom ≥50% of bone marrow nucleated cells are plasma cells (without transfusion support or thrombopoietin receptor agonist within 7 days before the laboratory test)

   - Absolute neutrophil count: ≥ 1.0×109/L (prior growth factor support is permitted but must be without support for 7 days for G-CSF or GM-CSF and for 14 days for pegylated GCSF before the laboratory test)

   - AST and ALT: ≤2.5×ULN
   * Creatinine clearance: ≥30 mL/min based on Cockcroft Gault equation
   * Total bilirubin: ≤2.0×ULN; except in participants with congenital bilirubinemia, such as Gilbert syndrome (in which case direct bilirubin ≤1.5×ULN is required)
   * Serum calcium corrected for albumin: ≤14 mg/dL (≤3.5 mmol/L) or free ionized calcium ≤6.5 mg/dL

   (ALT=alanine aminotransferase; AST=aspartate aminotransferase; GCSF=granulocyte colony stimulating factor; GM-CSF=granulocyte-macrophage colony stimulating factor; RBC=red blood cell; ULN=upper limit of normal)
9. A woman of childbearing potential must have a negative highly sensitive urine or serum (β human chorionic gonadotropin [β hCG]) pregnancy test at screening, again a negative serum test within 48 hours prior to the start of study treatment.
10. A woman must be:

    1. Not of childbearing potential, or
    2. Of childbearing potential and 1) Practicing true abstinence; or 2) Have a sole partner who is bilaterally vasectomized; or 3) Practicing 2 effective methods of contraception (at least 1 highly-effective, method of contraception (see 3 for methods of contraception allowed).

    NOTE: Participant must agree to continue the above throughout the study and for 100 days after the last dose of study treatment.

    NOTE: If a woman becomes of childbearing potential after start of the study the woman must comply with point (b) as described above. If a participant's reproductive status is questionable, additional evaluation should be considered.

    NOTE: An interaction between hormonal contraception and talquetamab has not been formally studied. Therefore, it is unknown whether talquetamab may reduce the efficacy of the contraception method. If a woman is receiving talquetamab and is using hormonal contraceptives, an additional barrier method must be used.

    NOTE: Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.
11. A woman must agree not to donate eggs (ova, oocytes) or freeze for future use, for the purposes of assisted reproduction during the study and for 100 days after receiving the last dose of study treatment
12. A man must wear a condom (with spermicidal foam/gel/film/cream/suppository) when engaging in any activity that allows for passage of ejaculate to another person during the study and for a minimum of 100 days after receiving the last dose of study treatment. If a female partner is of childbearing potential, she must also be practicing a highly effective method of contraception (see Section 13.2, Appendix 2).

    NOTE: If the male participant is vasectomized, he still must wear a condom (with foam/gel/film/cream/suppository), but his female partner is not required to use contraception.
13. A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 100 days after receiving the last dose of study treatment.
14. Must be willing and able to adhere to the lifestyle restrictions specified in this protocol ( Section 3.2), including to not donate blood or blood components during the study and for 100 days after the last dose of study drug). This includes complying with REMS program for lenalidomide. Per lenalidomide REMS program. In women of childbearing potential, pregnancy testing is needed weekly during the first month of treatment with lenalidomide, then monthly thereafter in females with regular menstrual cycles or every 2 weeks in females with irregular menstrual cycles.
15. Must sign an ICF (or their legally acceptable representative must sign) indicating that the participant understands the purpose of, and procedures required for, the study and is willing to participate in the study.
16. Willingness to return to study site for follow-up

Exclusion Criteria:

1. Intolerance to lenalidomide 10 mg (or 5 mg for patients with creatinine clearance 30-60 ml/min).
2. Refractory or relapsed multiple myeloma at any time before enrollment
3. Contraindications or life-threatening allergies, hypersensitivity, or intolerance to any study drug or its excipients (refer to the talquetamab Investigator's Brochure and appropriate package inserts).
4. Prior or concurrent exposure to any of the following, in the specified time frame as defined below:

   a. Received any prior GRPRCD5-directed therapy b. Received prior T-cell redirection therapy (for example, antibody therapy or BiTE's) or Chimeric antigen T cell therapy.

   b. Gene-modified adoptive cell therapy (eg, chimeric antigen receptor modified T cells, NK cells) within 3 months

   c. Targeted therapy, epigenetic therapy, or treatment with an investigational drug or an invasive investigational medical device within 21 days or ≥5 half-lives, whichever is less

   d. Investigational vaccine other than SARS CoV-2 vaccine approved/ in use under emergency approval within 4 weeks

   e. Live, attenuated vaccine within 4 weeks.

   f. Monoclonal antibody therapy targeting multiple myeloma within 21 days

   g. Cytotoxic therapy within 21 days i PI therapy within 14 days

   h. IMiD agent therapy within 14 days

   i. Radiotherapy within 14 days or focal radiation within 7 days
5. A maximum cumulative dose of corticosteroids of ≥ 140 mg of prednisone or equivalent within 14-day period before the first dose of study drug (does not include pretreatment medications) (Section 13.8, Appendix 8)
6. Known active CNS involvement or exhibits clinical signs of meningeal involvement of multiple myeloma. If either is suspected, negative whole brain MRI and lumbar cytology are required.
7. Plasma cell leukemia at the time of screening, Waldenström's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, M-protein, and skin changes), or primary amyloid light chain amyloidosis.
8. Myelodysplastic syndrome or active malignancies (ie, progressing or requiring treatment change in the last 24 months) other than relapsed/refractory multiple myeloma. The only allowed exceptions are:

   1. Non-muscle invasive bladder cancer treated within the last 24 months that is considered completely cured
   2. Skin cancer (non-melanoma or melanoma) treated within the last 24 months that is considered completely cured.
   3. Noninvasive cervical cancer treated within the last 24 months that is considered completely cured
   4. Localized prostate cancer (N0M0):

1. With a Gleason score of ≤7a, treated within the last 24 months, or untreated and under surveillance 2. With a Gleason score of 3+4 that has been treated >6 months prior to full study screening and considered to have a very low risk of recurrence, or e). History of localized prostate cancer and receiving androgen deprivation therapy and considered to have a very low risk of recurrence.

f) Breast cancer: adequately treated lobular carcinoma in situ or ductal carcinoma in situ, or history of localized breast cancer and receiving antihormonal agents and considered to have a very low risk of recurrence g) Other malignancy that is considered cured with minimal risk of recurrence.

9. Stroke, transient ischemic attack, or seizure within 6 months prior to signing ICF.

10. Participant is pregnant, breast-feeding, or planning to become pregnant while enrolled in this study or within 100 days after the last dose of study treatment.

11. Participant plans to father a child while enrolled in this study or within 100 days after the last dose of study treatment.

12. Presence of the following cardiac conditions:

1. New York Heart Association stage III or IV congestive heart failure
2. Myocardial infarction or coronary artery bypass graft ≤6 months prior to randomization
3. Uncontrolled cardiac arrhythmia or clinically significant ECG abnormalities
4. History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration
5. History of severe non-ischemic cardiomyopathy

   13. Any of the following:

a. Known to be seropositive for human immunodeficiency virus

1. Active hepatitis B infection (ie, HBsAg or HBV-DNA positive). In the event the infection status is unclear, quantitative viral levels are necessary to determine the infection status see Section 0 for further required assessments.
2. Active hepatitis C infection as measured by positive HCV-RNA testing. Participants with a history of HCV antibody positivity must undergo HCV-RNA testing. If a participant with history of chronic hepatitis C infection (defined as both HCV antibody and HCV-RNA positive) completed antiviral therapy and has undetectable HCV-RNA for at least 12 weeks following the completion of therapy, the participant is eligible for the study.

   14. Major surgery within 2 weeks prior to the start of administration of study treatment, or will not have fully recovered from surgery, or has major surgery planned during the time the participant is expected to be treated in the study or within 2 weeks after administration of the last dose of study treatment.

NOTE: Participants with planned surgical procedures to be conducted under local anesthesia may participate. Kyphoplasty or vertebroplasty are not considered major surgery. If there is a question whether a procedure is considered a major surgery, the investigator must consult with the study principal investigator and resolve any issues before enrolling a participant in the study.

15. Concurrent medical or psychiatric condition or disease that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study, such as:

1. Uncontrolled diabetes
2. Acute diffuse infiltrative pulmonary disease
3. Evidence of active systemic viral, fungal, or bacterial infection, requiring systemic antimicrobial therapy
4. Active autoimmune disease requiring systemic immunosuppressive therapy within 6 months before start of study treatment. EXCEPTION: Participants with vitiligo, controlled type I diabetes, and prior autoimmune thyroiditis that is currently euthyroid based on clinical symptoms and laboratory testing are eligible regardless of when these conditions were diagnosed.
5. Disabling psychiatric conditions (e.g., alcohol or drug abuse), severe dementia, or altered mental status
6. Any other issue that would impair the ability of the participant to receive or tolerate the planned treatment at the investigational site, to understand informed consent or any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

All subject files must include supporting documentation to confirm subject eligibility.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Stringent Complete Response (sCR) + Complete Response (CR) Rate | 12 months after the start of talquetamab in each participant.
  The primary outcome for this study, for the purposes of Clinical Trials.gov registration and results reporting, is the percentage of patients in complete response at 12 months.

SECONDARY OUTCOMES:
Minimal Residual Disease (MRD) negativity (10^-5) (ClonoSeqTM) | 2 years
  The percentage (%) of participants with MRD negativity (10^-5) (ClonoSeqTM) at 12 months after starting talquetamab.
Progression free survival (PFS) and overall survival (OS) | 4 years
  Percentage (%) of participants with PFS and OS up to 3 years after starting talquetamab.
Cytokine Release Syndrome (CRS), Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS), and hematologic and non-hematologic toxicities per NCI CTCAE v5 criteria | 1 year and 1 months post first patient treatment start
  Number of participants who experience a significant toxicity of interest (STI) in the first 3 months.
Quality of life - PROMIS® (Patient-Reported Outcomes Measurement Information System and Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE®) | 2 years
  PROMIS and PRO-CTCAE will be assessed monthly during study treatment and at end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Surbhi Sidana, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States